CLINICAL TRIAL: NCT00900549
Title: EvaluAtion of Resynchronization Therapy for Heart Failure (EARTH)
Brief Title: Evaluation of Resynchronization Therapy for Heart Failure
Acronym: EARTH
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Futility reason, no difference between study groups
Sponsor: Montreal Heart Institute (Other)
Collaborators: Abbott Medical Devices (Industry); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Bernard Thibault, MD, Montreal Heart Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCT67914 (Lesser Earth); ISRCTN 42560370
Record Dates: First submitted 2009-05-12; First posted 2009-05-13 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Heart Failure
Keywords: Heart failure; Cardiac resynchronization therapy; ICD
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CRT (Experimental)
  Interventions: Device: CRT on
- No CRT (Sham Comparator)
  Interventions: Device: CRT off

INTERVENTIONS:
Device: CRT on — 12 months
  Arms: CRT
Device: CRT off — 12-month
  Arms: No CRT

SUMMARY:
Heart failure is a major health problem in Canada. Recent advances in medical and device therapy have helped to reduce the morbidity and mortality of patients with this problem. Among these treatments, cardiac resynchronization therapy (CRT) has very recently been shown to be effective to improve functional class, quality of life and exercise tolerance of the patients with the most severe symptoms of heart failure and a prolonged duration of the QRS on the 12-lead Electrocardiography (ECG).

DETAILED DESCRIPTION:
Resynchronization of the failing ventricle is currently achieved by pacing the left and right ventricles simultaneously with specialized electrodes and a cardiac stimulator. However, controversy persists concerning the optimal configuration for cardiac pacing in these patients. Right ventricular pacing alone has been shown to be deleterious in some patient populations. The benefits of biventricular pacing in heart failure patients may be due primarily to left ventricular stimulation and may, in some patients, be decreased by the presence of simultaneous RV stimulation. Preliminary data from our own animal work suggest that in the majority of cases, LV stimulation alone is better than RV stimulation, and that BiV stimulation represents an intermediary situation between LV and RV stimulation.

ELIGIBILITY:
Inclusion Criteria:

* The patients are eligible if they undergo an ICD implantation or replacement
* They have a documented LVEF ≤ 35% measured in the previous 6 months (without major clinical subsequent event, such as heart surgery, since the LVEF measurement)
* If measured by echocardiography, the LV end-diastolic diameter must be ≥ 60 mm
* The duration of the QRS is < 120 ms
* They are in sinus rhythm
* They cannot walk more than 400 meters during the screening 6-minute walk test (the patients must be limited by heart failure symptoms)

Exclusion Criteria:

* Patients with an indication for permanent ventricular pacing or with chronotropic insufficiency defined as follow:

  * Any condition where the treating physician believes it would not be acceptable for the patient to have his device NOT programmed with the SENSOR at ON for the duration of the study
  * Second or third degree AV block, either persistent or intermittent
  * Patients with a pacemaker or an ICD who are paced in the ventricular chamber more than 5% of the time
* Patients with LV dysfunction associated with a reversible cause such as post-partum cardiomyopathy, tachycardia induced cardiomyopathy, acute myocarditis or acute toxic cardiomyopathy (including acute alcoholic)
* Patients who had a myocardial infarction within the past 6 weeks* defined by 2 of the 3 following conditions:

  * Prolonged chest pain
  * ECG changes suggesting of AMI
  * Cardiac enzymes elevation more than twice the local upper limit of normal)
* Patients who had cardiac surgery within the past 6 weeks*
* Patients with moderate or severe cardiac valve stenosis (aortic, mitral, pulmonary or tricuspid)
* Patients with an inability or a limitation to walk for reasons other than heart failure symptoms (e.g., angina, intermittent claudication, severe lung condition or arthrosis)
* Patients with severe coexisting illnesses making survival > 6 months unlikely
* Patients who are pregnant and/or nursing.
* Patients with inability or unwillingness to consent or comply with follow-up requirements
* Patients participating in another study

The 6-week period is calculated prior to the beginning of the baseline evaluation and not the implant procedure itself. This difference comes from the fact that the protocol includes a delay of 2 to 8 weeks between the implant procedure and the actual beginning of the patient's evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2003-10; Primary Completion 2011-02 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Total exercise duration at a constant submaximal load (defined as 75% of peak exercise during the baseline metabolic evaluation); study is powered to detect a min difference of 300 sec (+25% from baseline) in the primary endpoint between the 2 treatments | one year

SECONDARY OUTCOMES:
Clinical & electrical endpoints and echocardiographic & nuclear medicine evaluation of LV function. Dyssynchrony evaluation will help advancing the understanding of the physiopathology of heart failure and response to resynchronization therapy. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Thibault, MD, Study Chair — Montreal Heart Institute
Locations (11):
- Canada (11):
  - University of Alberta Hospital, Edmonton, Alberta
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences Center, Hamilton, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Sunnybrook & Women's Hospital, Toronto, Ontario
  - St-Michael's Hospital, Toronto, Ontario
  - CHUS-Fleurimont, Fleurimont, Quebec
  - CHUM-Hôpital Hotel-Dieu, Montreal, Quebec
  - Sacre-Coeur Hospital, Montreal, Quebec
  - Montreal Heart Institute Research Center, Montreal, Quebec
  - Institut Univ de Cardiologie et de Pneumologie de Québec, Québec, Quebec

REFERENCES:
- [Derived] Thibault B, Harel F, Ducharme A, White M, Ellenbogen KA, Frasure-Smith N, Roy D, Philippon F, Dorian P, Talajic M, Dubuc M, Guerra PG, Macle L, Rivard L, Andrade J, Khairy P; LESSER-EARTH Investigators. Cardiac resynchronization therapy in patients with heart failure and a QRS complex <120 milliseconds: the Evaluation of Resynchronization Therapy for Heart Failure (LESSER-EARTH) trial. Circulation. 2013 Feb 26;127(8):873-81. doi: 10.1161/CIRCULATIONAHA.112.001239. Epub 2013 Feb 6. PMID 23388213